CLINICAL TRIAL: NCT06969534
Title: Phase II Clinical Study on the Safety and Efficacy of Pucotenlimab Combined With the Chemotherapy Regimen of Gemcitabine and Cisplatin for Lymphoepithelioma-like Carcinoma in Children and Adolescents
Brief Title: Safety and Efficacy of Pucotenlimab in pLECC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhuo Zhang, Director of department of pediatric cancer,Principal Investigator,Clinical Professor,, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLECC-1001
Record Dates: First submitted 2025-04-23; First posted 2025-05-14 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Lymphoepithelioma-like Carcinoma; Lymphoepithelioma; Carcinoma
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pucotenlimab plus a fixed regimen( Gemcitabine and cisplatin) (Experimental)
  Interventions: Drug: Pucotenlimab combined with GP regimen

INTERVENTIONS:
Drug: Pucotenlimab combined with GP regimen — A total of 33 cases are planned to be enrolled. All the subjects will receive Pucotenlimab (3mg/kg, on day 1, with a maximum dose not exceeding 200mg), administered once every 3 weeks (Q3W), and combined with the GP regimen. The chemotherapy is a fixed regimen, with Gemcitabine at a dose of 1g/m² on day 1 and day 8, and cisplatin at a dose of 80mg/m² on day 1. The chemotherapy will be given for 3 to 6 cycles, once every 3 weeks (Q3W).

SUMMARY:
Lymphoepithelioma-like carcinoma (LELC) in children is a rare epithelial malignant tumor. Regarding pediatric lymphoepithelioma-like carcinoma (pLELC), its clinicopathological features, prognosis, and molecular characteristics remain unknown. In preclinical studies, this study aims to explore the safety and efficacy of the PD-1 monoclonal antibody pucotenlimab combined with the chemotherapy regimen of gemcitabine and cisplatin as the first-line treatment for lymphoepithelioma-like carcinoma in children and adolescents.

DETAILED DESCRIPTION:
Lymphoepithelioma-like carcinoma (LELC) in children is a rare epithelial malignant tumor, and its most prominent feature is the presence of a large number of tumor infiltrating lymphocytes (TILs) in the tumor background. LELC can occur in various organs of the digestive, respiratory, skin, urinary, reproductive and other systems, but it is most commonly found in the lungs, salivary glands and stomach. In children, the common sites of LELC are the thymus, parotid gland, lymph nodes and other parts. Clinically, there is no standard treatment guideline for LELC, and currently, the same treatment regimens as those for other tumors in the same system are mostly used. At present, there is a lack of systematic reports on pediatric lymphoepithelioma-like carcinoma (pLELC), and most of the known reports are case studies.

For pediatric lymphoepithelioma-like carcinoma (pLELC), its clinicopathological features, prognosis and molecular characteristics remain unknown. Previously published research of the investigators showed that in preclinical studies, the clinical features and prognosis of pLELC were reported, and a retrospective study explored the real-world efficacy data of the investigators' center over more than 10 years. Kaplan-Meier survival analysis for children and adolescents showed that for patients who only received chemotherapy, the 1-year progression-free survival (PFS) was 60.72% (95% CI: 45.07% - 81.79%), and the 2-year progression-free survival was 56.92% (95% CI: 41.18% - 78.68%). The 1-year overall survival (OS) of the patients was 96.4% (95% CI: 89.79% - 100%), and the 2-year overall survival was 76.53% (95% CI: 61.66% - 95.00%).

For the group treated with PD-1 inhibitor combined with chemotherapy, only 1 patient (1/10) died due to disease progression. Kaplan-Meier survival analysis showed that for patients who received anti-PD-1 combined with chemotherapy, the 1-year progression-free survival was 100%, and the 2-year progression-free survival was 72.92% (95% CI: 46.80% - 100%). In addition, the 1-year overall survival of patients who received anti-PD-1 combined with chemotherapy was 100%, and the 2-year overall survival was 87.5% (95% CI: 67.34% - 100%). Both the median progression-free survival and the median overall survival have not been reached.

In addition, the investigators determined its genomic landscape through whole exome sequencing (WES), including single nucleotide variants (SNVs) and copy number variants (CNVs). Furthermore, the investigators comprehensively compared the genomic landscape of pLELC with other related cancer types (such as nasopharyngeal carcinoma in children and adult LELC) to further deepen understanding of this malignant tumor.

The preclinical data provide a theoretical basis for the immunotherapy with PD-1 antibody for pediatric lymphoepithelioma-like carcinoma.

This study aims to explore the safety and efficacy of the PD-1 monoclonal antibody pucotenlimab combined with the chemotherapy regimen of gemcitabine and cisplatin as the first-line treatment for lymphoepithelioma-like carcinoma in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Age: Between 1 and 18 years old;
* ECOG PS score: 0 to 1 point;
* Histopathologically confirmed locally advanced or metastatic lymphoepithelioma-like carcinoma in children or adolescents;
* Must have at least one measurable lesion defined by the RECIST or WHO criteria;
* Estimated survival time ≥ 6 months;
* Cardiac function:Left ventricular ejection fraction (LVEF) detected by echocardiography ≥ 50%; Electrocardiogram (EKG) shows no signs of myocardial ischemia;
* No history of arrhythmia requiring drug intervention before enrollment;
* No history of severe immune-related adverse events (CTCAE V4.03 Grade 3 or Grade 4);
* For patients known not to have bone marrow (BM) involvement:Absolute neutrophil count (ANC) ≥ 1.0×10⁹/L; Platelet count ≥ 100.0×10⁹/L;Hemoglobin ≥ 90 g/L;
* Liver and kidney functions should meet the following criteria: Total bilirubin (conjugated + unconjugated) ≤ 2.5× the upper limit of normal value (ULN) (corresponding to the age). Patients with confirmed Gilbert's syndrome can be considered for enrollment at the discretion of the investigator;Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5× ULN; Estimated glomerular filtration rate ≥ 30 mL/min/1.73 m² or serum creatinine (Cr) ≤ 1.5× ULN;
* During participation in the study, be able to comply with outpatient treatment, laboratory monitoring and necessary clinical visits;
* The parents/guardians of child or adolescent subjects are capable of understanding, consenting to and signing the Informed Consent Form (ICF) for the study and the applicable child consent form before any protocol-related procedures are initiated. With the consent of the parents/guardians, the subject is capable of expressing consent (when applicable).

Exclusion Criteria:

* Have received anti-PD-1 or anti-PD-L1 monoclonal antibodies or targeted drugs of related pathways;
* Known to be allergic to PD-1 monoclonal antibody or any of its excipients; Known to have a history of allergic diseases or have a severe allergic constitution;
* Have other malignant tumor diseases other than the tumor being treated in this study, except for: Malignant tumors that have been cured and have not recurred within 3 years before study enrollment, completely resected basal cell and squamous cell skin cancers, and any type of in-situ cancer that has been completely resected;
* Active central nervous system metastases (whether treated or not), including symptomatic brain metastases, meningeal metastases, spinal cord compression, etc.; Except for: Asymptomatic brain metastases (no progression within at least 4 weeks after radiotherapy and/or no neurological symptoms or signs after surgical resection, and no need for dexamethasone or mannitol treatment).
* Uncontrollable pleural effusion, pericardial effusion or ascites that requires repeated drainage;
* The toxicity of previous treatment is still > Grade 1 (CTCAE V4.03 criteria), except for alopecia and neurotoxicity;
* Have a history of mental disorders;
* Have a history of drug abuse or drug addiction as determined by inquiry;
* Have a history of idiopathic pulmonary fibrosis or idiopathic pneumonia;
* Have comorbidities that require treatment with immunosuppressive drugs, or have comorbidities that require systemic or local use of corticosteroids at immunosuppressive doses (prednisone > 10 mg/day or equivalent dose of similar drugs).
* Have a history of autoimmune diseases, including but not limited to systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory bowel disease, Hashimoto's thyroiditis, etc., except for: Type 1 diabetes mellitus, hypothyroidism that can be controlled only by hormone replacement therapy, skin diseases that do not require systemic treatment (such as vitiligo, psoriasis), celiac disease that has been controlled, or diseases that are not expected to recur without external stimulating factors;
* Have a history of previous or current active tuberculosis infection;
* Have active infections that require systemic treatment;
* Uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg), or pulmonary hypertension, or unstable angina pectoris; Have had a myocardial infarction or undergone coronary artery bypass grafting or stenting surgery within 6 months before drug administration; Have a history of chronic heart failure meeting New York Heart Association (NYHA) criteria Class 3-4; Have clinically significant valvular heart disease; Have severe arrhythmias that require treatment (excluding atrial fibrillation and paroxysmal supraventricular tachycardia), including a QTc interval of ≥ 450 ms for men and ≥ 470 ms for women (calculated by the Fridericia formula); Have had a cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months before drug administration, etc.;
* Have severe medical comorbidities, including but not limited to: Uncontrolled diabetes mellitus, active peptic ulcer, active bleeding, etc.;
* Positive for Anti-HIV, TP-Ab, HCV-Ab; Positive for HBV-Ag and the HBV DNA copy number > the upper limit of the normal value of the testing unit;
* Abnormal thyroid function test results (FT3, FT4, T3, T4);
* Expected to receive live vaccines or attenuated vaccines within 4 weeks before drug administration, during the treatment period, or within 5 months after the last drug administration;
* Have participated in another clinical trial and received the investigational drug treatment within 30 days before drug administration;
* Patients who, according to the judgment of the investigator, are not suitable for participating in this trial for other reasons.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | PFS is defined as the time interval from the start of treatment until the occurrence of disease progression or death of the patient from any cause, whichever happens first (up to 24 months）.
  progression of the disease or the death

SECONDARY OUTCOMES:
ORR | The objective response rate will be assessed over an estimated period of up to 3 months（after first 2 cycles, before the 3rd cycle, each cycle is 21 days).
  The objective response rate is an important indicator for measuring the effect of a treatment regimen in shrinking tumors.Starting from the initiation of the combination therapy, regular imaging examinations (such as CT, MRI, etc.) and clinical evaluations of patients will be conducted.
OS | The assessment of OS will be carried out over an estimated period of up to 24 months.
  Overall survival (OS) is defined as the time from the initiation of treatment with pucotenlimab in combination with the GP regimen until the patient's death from any cause. Death is determined based on official medical records or other reliable documentation. The follow - up for OS will continue throughout this estimated assessment period.

CONTACTS AND LOCATIONS:
Locations (1):
- Yizhuo Zhang, Guangzhou, Guangdong, China